CLINICAL TRIAL: NCT04602260
Title: Functional Recovery of Older Hospitalised Patients With COVID-19: a Prospective and Retrospective Cohort Study Extension to the Coronavirus Registry (COREG)
Brief Title: Functional Recovery of Hospitalised Patients With COVID-19: The COREG Extension Study
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Marla Beauchamp, Assistant Professor, McMaster University
Other Study IDs: COREG-Extension_14567
Record Dates: First submitted 2020-09-03; First posted 2020-10-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Covid19; Corona Virus Infection; Mobility Limitation; Frailty
Keywords: mobility; functional recovery; pulmonary function; Covid-19; coronavirus; health outcomes
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Mobility Limitation; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: The prospective cohort will assess patients upon admission to general internal medicine, at hospital discharge, and at 3, 6, 9, and 12-month follow-up.
- Retrospective Cohort: The retrospective cohort will assess patients at 3, 6, 9, and 12-months after being discharged from the hospital.

SUMMARY:
Older adults and those with chronic underlying health conditions are the most susceptible to COVID-19 and its complications. Although there has been a rapid response to studying the effects of COVID-19 in the acute stages, little is known about recovery over the longer-term. Older adults who survive the diseases are at risk of developing persistent mobility limitations due to extensive bed rest during hospitalization. For older patients and those with underlying frailty recovering from COVID-19, this could rapidly lead to significant physical deconditioning and rapid declines in mobility. Understanding the trajectory of functional recovery of older hospitalised patients with COVID-19 in the short- and long-term is critical to improving patient outcomes and informing health and rehabilitative interventions for survivors.

DETAILED DESCRIPTION:
The coronavirus disease of 2019 (COVID-19) is an international public health challenge with far-reaching social, economic and health impacts. Older adults and those with chronic underlying health conditions are the most susceptible to COVID-19 and its complications. Of the 15,381 reported cases of COVID-19 in Ontario to date, approximately 22.2% (n=3,420) are aged 60-79 and 22.4% (n=3,443) are 80 and over. Although there has been a rapid and coordinated response to studying the effects of COVID-19 in the acute stages, little is known about recovery over the longer-term. Anecdotally, the investigators are seeing severe declines in function, persistent symptoms, and new and worsening chronic conditions among older survivors of COVID-19. It is known that older adults who survive acute respiratory distress syndrome and associated diseases are at risk of developing persistent mobility limitations due to extensive bed rest and/or long stays in the intensive care unit (ICU) during hospitalization. Recent studies have shown that many older patients spend only 4% of their hospital stay out of bed, and each day in bed is associated with a 1-5% loss in muscle strength. For older patients and those with underlying frailty recovering from COVID-19, this could rapidly lead to significant physical deconditioning and rapid declines in mobility; with further losses in physiological reserve and resilience. Understanding the trajectory of functional recovery of older hospitalised patients with COVID-19 in the short- and long-term is critical to improving patient outcomes and informing health and rehabilitative interventions for survivors.

This study is an extension of the Coronavirus (COVID-19) Registry (COREG) platform (PI Andrew Costa)- a unique Kitchener-Waterloo-Hamilton registry of suspected and confirmed COVID-19 hospital admissions based on (and in collaboration with) the WHO International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC). The addition of a prospective cohort study extension to COREG will allow the investigators to follow-older hospitalised COVID-19 patients over the longer-term in order to gain an understanding of the trajectory of functional recovery of the disease. Combining the primary data collection with COREG will also allow the investigators to identify determinants of long-term outcomes for at-risk older adults. These data are necessary to guide the clinical care and optimal management of older patients who survive serious COVID-19 illness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently hospitalised/recently discharged due to/since confirmed or suspected COVID- 19 infection using the ISARIC definition.

Exclusion Criteria:

* Previously institutionalized
* Pre-morbid severe mobility limitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients included in the COREG registry that meet inclusion criteria will be approached for enrollment in this extension study.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Activity Measure for Post Acute Care (AM-PAC) Basic Mobility Inpatient Version | Admission to hospital ward (0-14 days post ward admission) and discharge from hospital (0-14 days post discharge or up to 6 months, whichever comes first)
  The AM-PAC is an activity limitation instrument based on the International Classification of Functioning, Disability and Health (ICF) that assesses 3 functional domains: basic mobility, daily activities and applied cognition.
Change in Activity Measure for Post Acute Care (AM-PAC) Basic Mobility Outpatient Version | Admission to hospital ward (0-14 days post ward admission, to capture pre-morbid function), and at 3,6,9 and 12-months post hospital discharge
  The AM-PAC is an activity limitation instrument based on the International Classification of Functioning, Disability and Health (ICF) that assesses 3 functional domains: basic mobility, daily activities and applied cognition.
Change in Activity Measure for Post Acute Care (AM-PAC) Applied Cognitive Inpatient Version | Admission to hospital ward (0-14 days post ward admission) and discharge from hospital (0-14 days post discharge or up to 6 months, whichever comes first)
  The AM-PAC is an activity limitation instrument based on the International Classification of Functioning, Disability and Health (ICF) that assesses 3 functional domains: basic mobility, daily activities and applied cognition.
Change in Activity Measure for Post Acute Care (AM-PAC) Daily Activity | 3,6,9 and 12-months post hospital discharge
  The AM-PAC is an activity limitation instrument based on the International Classification of Functioning, Disability and Health (ICF) that assesses 3 functional domains: basic mobility, daily activities and applied cognition.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) | 3,6,9 and 12-months post hospital discharge
  The SPPB combines the results of gait speed over 3 meters, the 5-repetition chair-stand, and a progressive balance test to assess lower extremity function.
Change in Clinical Frailty Scale (CFS) for participants over 60 years of age | Admission to hospital ward (0-14 days post ward admission, to capture pre-morbid function ), and at 3,6,9 and 12-months post hospital discharge
  The CFS is an interview-based scale wherein the assessor may ask the participant questions about things such as a participant's independence or physical abilities to determine where the participant falls along the 9-point scale, from 1 (Very Fit) to 9 (Terminally Ill).
Change in Forced Expiratory Volume (FEV1) | 3,6,9 and 12-months post hospital discharge
  The Forced Expiratory Volume in 1 Second parameter measures the volume of air that was exhaled into the mouthpiece in the first second after a full inhalation as measured by spirometry.
Change in Forced Vital Capacity (FVC) | 3,6,9 and 12-months post hospital discharge
  The amount of air that can be forcibly exhaled from a participant's lungs after taking the deepest breath possible, as measured by spirometry. FVC is the total amount of air exhaled during the FEV test.
Change in Forced Expiratory Volume Percentage (FEV1%) | 3,6,9 and 12-months post hospital discharge
  The FEV1/FVC Ratio (FEV1%) parameter is calculated by dividing the measured FEV1 value by the measured FVC value.
Change in Functional Independence Measure (FIM) | 3 and 6 months post hospital discharge
  The FIM assesses the functional status of a person based on the level of assistance the person requires.
Change in Impact of Event Scale - Revised (IES-R) | 3,6,9 and 12-months post hospital discharge
  The IES-R is a 22-item self-report measure that asks questions about subjective distress caused by traumatic events. Each item is rated on a 5-point scale, from 0 ("not at all") to 4 ("extremely").
Change in Health status (EQ-5D-5L) | 3,6,9 and 12-months post hospital discharge
  The EQ-5D-5L is a generic and well-established instrument for describing health status or disease-specific outcome measures. It defines health in terms of five dimensions: Mobility, Self- Care, Usual Activities, Pain/Discomfort, and Anxiety/ Depression. The response options are of five levels, from no, slight, moderate, severe, to extreme problems
Change in Post-COVID-19 Functional Status Scale (PCFSS) | 3,6,9 and 12-months post hospital discharge
  Developed in early 2020, this 5-point scale assesses how individuals have been affected in a participant's everyday life by COVID-19 illness and recovery. Lower grades indicate better functioning, with grade 0 representing the absence of symptoms or functional limitations and grade 4 reflecting severe limitations and symptom burden. The PCFSS can be patient-reported following a flow diagram series of questions to result in a grade, or it can be administered via structured interview, which is more comprehensive. The research team will conduct the structured interview over the phone and the patient-reported flow chart during the home visits.
Change in Hospital Anxiety and Depression Scale (HADS) | 3,6,9 and 12-months post hospital discharge
  The HADS is a 14-item two-dimension scale that identifies depression and anxiety among physically ill patients. Scores range from 0 to 21, with higher scores indicating higher levels of anxiety. In the general ill population, a cut-off of ≥8 indicates depression.
Change in Fatigue Visual Analog Scale (Fatigue VAS) | 3,6,9 and 12-months post hospital discharge
  This visual scale allows individuals to rate a participant's global fatigue from 0 (worst fatigue) to 10 (normal).
Change in Modified Medical Research Council (MRC) Breathlessness Scale | 3,6,9 and 12-months post hospital discharge
  This brief questionnaire contains five statements describing a range of breathlessness from only becoming breathless with strenuous exercise to being too breathless to leave the house.
Change in Oxygen Saturation (SpO2) | 3,6,9 and 12-months post hospital discharge
  Oxygen saturation will be measured using a fingertip pulse oximeter to detect hypoxia and to evaluate any persistent hypoxia post-COVID-19 illness.

CONTACTS AND LOCATIONS:
Overall Officials: Marla K Beauchamp, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reid JC, Costa AP, Duong M, Ho T, Kruisselbrink R, Raina P, Kirkwood R, Jones A, Corriveau S, Griffith LE, Haider S, Marcucci M, Markle-Reid M, Morrison H, Raghavan N, Schumacher C, Vrkljan B, Junek M, Martin L, Patel A, Girolametto C, Pitre T, Beauchamp MK; COREG Investigators. Functional recovery following hospitalisation of patients diagnosed with COVID-19: a protocol for a longitudinal cohort study. BMJ Open. 2021 Dec 13;11(12):e053021. doi: 10.1136/bmjopen-2021-053021. PMID 34903545
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343